CLINICAL TRIAL: NCT06285487
Title: Depression in Youth Onset Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1600
Record Dates: First submitted 2024-02-15; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes; Depression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpersonal Psychotherapy adapted for Type 2 Diabetes (Experimental): Participants in the IPT-T2D will receive 1 hour weekly IPT from a licensed psychologist in a group setting for 6 weeks.
  Interventions: Behavioral: Group Program
- Health Education adapted for Type 2 Diabetes (Experimental): Participants in the Health Education-T2D will receive 1 hour weekly Health Education lessons from a licensed psychologist in a group setting for 6 weeks.
  Interventions: Behavioral: Group Program

INTERVENTIONS:
Behavioral: Group Program — Participants in both arms will receive 6 weeks of T2D-IPT or 6 weeks of T2DEd.

SUMMARY:
The main purpose of this study is to compare a group-based interpersonal psychotherapy (IPT) program and a Type 2 Diabetes education program to determine if there are differences in depression levels, diabetes distress, and glycemic control in adolescents with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes diagnosis ≥ 3 months
* Age 12-17yr
* Elevated depression symptoms
* HbA1c ≥7.0%

Exclusion Criteria:

* Currently receiving psychotherapy from a licensed counselor
* Psychotropic meds <8 weeks

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability of IPT-T2D | 3 Months
  Assessed by likeability, credibility, and descriptions by adolescents, parents, and facilitators
Depression Changes | 3 Months
  Assessed by CESD
Changes in Glycemic Control | 3 Months
  Assessed by changes in HbA1c

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States